CLINICAL TRIAL: NCT00765492
Title: A Phase I, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD8529 When Given as Single and Multiple Ascending Oral Doses in Healthy Subjects
Brief Title: AZD8529 Multiple Ascending Dose Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark A. Smith, MD; Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: D1960C00002
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2009-06-26 (Estimated); Status verified 2009-06

CONDITIONS: Healthy Volunteer
Keywords: Phase I
MeSH Terms: interventions — AZD8529

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD8529
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8529 — oral
  Arms: 1
Drug: Placebo — oral
  Arms: 2

SUMMARY:
This is a study to evaluate safety, tolerability, PK and PD effects of orally administered AZD8529 after multiple ascending doses

ELIGIBILITY:
Inclusion Criteria:

* Female subjects must be of non-child bearing potential.

Exclusion Criteria:

* Has received another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment within 30months of the first administration of investigational prod
* Plasma donation within one month of screening or any blood donation/blood loss > 500mL during the 3 months prior to screening
* Clinically relevant abnormalities in physical examinations, vital signs, ECG, clinical chemistry, hematology or urinalysis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Estimated)
Dates: Start 2008-10; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of multiple dose administration of AZD8529 when given orally to healthy male subjects and female subjects of non-childbearing potential. | each visit, at least daily, during the study.

SECONDARY OUTCOMES:
To characterize the pharmacokinetics of AZD8529 in plasma | Blood samples will be taken during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Smith, MD, PhD, Study Director — AstraZeneca